CLINICAL TRIAL: NCT07174102
Title: Radiologic Features of Patients With Rheumatoid Arthritis Related Interstitial Lung Disease at Chest High Resolution Computed Tomography
Brief Title: Radiologic Features of Rheumatoid Arthritis Interstitial Lung Disease at Chest High Resolution Computed Tomography
Status: Recruiting | Type: Observational
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Collaborators: University of Parma (Other)
Responsible Party: Sponsor
Other Study IDs: ARD-ILD-HRCT
Record Dates: First submitted 2025-08-14; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Reumatoid Arthritis; Interstitial Lung Disease Due to Systemic Disease (Disorder); Idiopathic Pulmonary Fibrosis (IPF); Connective Tissue Disease (CTD)
Keywords: rheumatoid arthritis; Interstitial lung disease; connective tissue disease; idiopathic pulmonary fibrosis; high resolution computed tomography
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Connective Tissue Diseases; Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rheumatoid arthritis-interstitial lung disease group: Patients with rheumatoid arthritis related interstitial lung disease undergoing to HRCT at any time of their clinical history
  Interventions: Diagnostic Test: High resolution computed tomography
- Idiopathic pulmonary fibrosis: Patients with idiopathic pulmonary fibrosis underoging to HRCT at any time of their clincial history
  Interventions: Diagnostic Test: High resolution computed tomography
- Connective tissue disease - interstitial lung disease: Patients with connective tissue diseases related interstitial lung disease undergoing to HRCT at any time of their clinical history
  Interventions: Diagnostic Test: High resolution computed tomography

INTERVENTIONS:
Diagnostic Test: High resolution computed tomography — High resolution computed tomography perfomed in patients with rheumatoid arthritis and connective tissue diseases with or without interstitial lung disease, and idiopathic pulmonary fibrosis

SUMMARY:
Lung involvement is one of the most frequent extra articular involvements of rheumatoid arthritis (RA). RA related lung involvement can affect parenchyma, airway, vascular tree and serosa. Among all possible manifestations of lung disease, interstitial lung disease is the most severe being able to compromise quality of life and survival and involves about 20% of patients with rheumatoid arthritis (RA). However, chest high resolution computed tomography (HRCT) features of RA, with or without interstitial lung involvement, have not been clearly defined. Such features have been mostly investigated on small populations of RA patients, often including patients with connective tissue diseases (CTDs), namely systemic sclerosis, mixed connective tissue disease, idiopathic inflammatory myopathies, making difficult to discriminate possible specific features of RA interstitial lung disease (ILD).

The aims of this observational longitudinal study are to investigate: i) chest HRCT features of RA (frequency of radiologic HRCT patterns, fibrosis, nodules, bronchiectasis, etc.), associated or not to ILD; ii) possible associations between chest HRCT features and demographic, clinical and serologic characteristics of RA; iii) specific chest HRCT features of RA ILD, compared to idiopathic pulmonary fibrosis (IPF) and CTD ILD (i.e., primary Sjogren syndrome, idiopathic inflammatory myopathies, etc), according to the Centres availability.

Consecutive, unselected, DICOM files of chest HRCT of adult RA patients (regardless a previous diagnosis of ILD) will be evaluated by an expert thoracic radiologist blinded to patients' clinical history.

HRCT patterns, presence of fibrosis and other lung abnormalities (cysts, nodules, pleural effusion, etc) will be recorded. In patients with RA ILD possible associations with demographic and clinical disease features will be also analysed (such as sex, disease duration, disease duration at ILD diagnosis, presence of ACPA, rheumatoid factor, ANA), inclusion of previous therapies.

After 2 years, new HRCT and lung function tests will be collected for each enrolled patients when available, to evaluate possible changes of lung involvement over time.

DETAILED DESCRIPTION:
Lung involvement is one of the most frequent extra-articular involvements of rheumatoid arthritis (RA). RA-related lung involvement can affect parenchyma, airway, vascular tree and serosa. Among all possible manifestations of lung disease, interstitial lung disease is the most severe being able to compromise quality of life and survival and involves about 20% of patients with rheumatoid arthritis (RA).

However, chest high resolution computed tomography (HRCT) features of RA, with or without interstitial lung involvement, have not been clearly defined. Such features have been mostly investigated on small populations of RA patients, often including patients with connective tissue diseases (CTDs), namely systemic sclerosis, mixed connective tissue disease, idiopathic inflammatory myopathies, making difficult to discriminate possible specific features of RA-interstitial lung disease (ILD).

This observational longitudinal study aims to investigate:

* Chest HRCT features of RA-ILD (frequency of radiologic HRCT patterns, fibrosis, nodules, bronchiectasis, etc). Possible findings specific for RA independently from ILD will be also analysed.
* Possible associations between chest HRCT features and demographic, clinical and serologic characteristics of RA.
* Specific chest HRCT features of RA-ILD, compared to idiopathic pulmonary fibrosis (IPF) and CTD-ILD (i.e., primary Sjogren syndrome, idiopathic inflammatory myopathies, etc) according to the Centres availability.

All consecutive RA patients, older than 18 and able to understand the aims of the study and undergoing HRCT for clinical needs will be enrolled in the study.

Patients with idiopathic pulmonary fibrosis and other CTDs undergoing to HRCT will be enrolled as control groups Patients younger than 18 and unable to give their informed consent will be excluded from the study

Consecutive, unselected, DICOM files of chest HRCT of RA patients (regardless a previous diagnosis of ILD) will be evaluated by an expert thoracic radiologist blinded to patients' clinical history. The DICOM images will be anonymized, coded and sent to the coordinating centre by transfer to a dedicated server whose access will be protected by a password. If deemed clinically necessary, patients will also be evaluated by a pulmonologist expert in the treatment of fibrosing lung diseases.

HRCT patterns, presence of fibrosis and other lung abnormalities (cysts, nodules, pleural effusion, etc) will be recorded. In patients with RA-ILD possible associations with demographic and clinical disease features will be also analysed (such as sex, disease duration, disease duration at ILD diagnosis, presence of ACPA, rheumatoid factor, ANA), inclusion of previous therapies.

RA diagnosis must be performed according to 2010 EULAR/ACR classification criteria, overlap syndrome are excluded from the study.

To evaluate specific HRCT features of RA-ILD, consecutive, unselected DICOM files of chest HRCT of patients with IPF and CTD-ILD (i.e., primary Sjogren syndrome, idiopathic inflammatory myopathies or other, according to the Centres availability) will be also evaluated by an expert thoracic radiologist blinded to patients' clinical history.

After 2 years, new HRCT and lung function tests will be collected for each enrolled patients when available, to evaluate possible changes of lung involvement over time.

ELIGIBILITY:
Inclusion Criteria:

* patients able to give their informed consent
* at least aged 18 years
* patients undergoing High-Resolution Computed Tomography (HRCT) for clinical needs at any point in their medical history
* patients with a diagnosis of rheumatoid arthritis, idiopathic pulmonary fibrosis or connective tissue disease

Exclusion criteria:

Patients younger than 18 and unable to give their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients or with idiopathic pulmonary fibrosis and other connective tissue diseases
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of radiologic interstitial lung disease patterns | At baseline and 24 months
  Prevalence of radiologic interstitial lung disease patterns in patients with rheumatoid arthritis related interstitial lung disease compared with other rheumatic diseases
Prevalence of honeycombing | At baseline and 24 months
  Prevalence of honeycombing in rheumatoid arthritis patients related interstitial lung disease compared to other rheumatic diseases at the enrollment
Prevalence of anterior honeycombing | At baseline and 24 months
  Prevalence of anterior honeycombing in patients with rheumatoid related interstitial lung disease compared with other rheumatic diseases and idiopatic pulmonary fibrosis
Progression of fibrotic features | At baseline and 24 months
  New HRCT will be collected for each enrolled patients when available, to evaluate possible changes of fibrotic features described at baseline

SECONDARY OUTCOMES:
Prevalence of exuberant honeycombing | At baseline and 24 months
  Prevalence of exuberant honeycombing in patients with rheumatoid related interstitial lung disease compared with other rheumatic diseases and idiopatic pulmonary fibrosis
Prevalence of straight sign | At baseline and 24 months
  Prevalence of exuberant honeycombing in patients with rheumatoid related interstitial lung disease compared with other rheumatic diseases and idiopatic pulmonary fibrosis

CONTACTS AND LOCATIONS:
Locations (5):
- Institute of Rheumatology, Na Slupi 4, Prague, Czechia
- Italy (4):
  - UOC Reumatologia, Arcipedale Sant'Anna, Ferrara
  - SC Malattie Apparato Respiratorio, Azienda Policlinico di Modena, Modena
  - Local Health Unit ("Azienda Unità Sanitaria Locale", AUSL) of Piacenza, Piacenza
  - AUSL-IRCCS di Reggio Emilia, Reggio Emilia